CLINICAL TRIAL: NCT05898672
Title: A PHASE 1, RANDOMIZED, FIXED SEQUENCE, MULTIPLE-DOSE, OPEN-LABEL STUDY TO ESTIMATE THE EFFECT OF NIRMATRELVIR (PF-07321332)/RITONAVIR ON ROSUVASTATIN PHARMACOKINETICS IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn About the Study Medicine Called Nirmatrelvir/Ritonavir in People Who Are Healthy Volunteers Co-administered the Medicine Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C4671052; 2023-503570-20 (EudraCT Number: CTIS (EU)); 2023-503570-20-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Pharmacokinetics; Healthy Volunteers
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Nirmatrelvir; Paxlovid; Rosuvastatin
MeSH Terms: conditions — COVID-19 | interventions — Rosuvastatin Calcium; nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A: rosuvastatin (Active Comparator): Rosuvastatin tablets
  Interventions: Drug: Rosuvastatin
- Treatment B: rosuvastatin + nirmatrelvir/ritonavir (Experimental): Rosuvastatin + nirmatrelvir/ritonavir tablets
  Interventions: Drug: Rosuvastatin; Drug: Nirmatrelvir/ritonavir

INTERVENTIONS:
Drug: Rosuvastatin — Single oral dose of rosuvastatin tablets
Drug: Nirmatrelvir/ritonavir — Twice daily oral doses of nirmatrelvir/ritonavir tablets
  Arms: Treatment B: rosuvastatin + nirmatrelvir/ritonavir

SUMMARY:
The purpose of this study is to learn about the effect of the study medicine (called nirmatrelvir/ritonavir) on the pharmacokinetics of the medicine rosuvastatin in healthy volunteers. Pharmacokinetics helps us understand how the drug is changed and eliminated from your body after you take it.

This study is seeking participants who:

* are male and female participants who are overtly healthy
* are 18 years of age or older
* have a Body mass Index (BMI) of 16-32 kg/m2 and total body weight >50 kg (110 lb).

All participants in this study will receive nirmatrelvir/ritonavir, a standard treatment for mild-to-moderate COVID-19. All participants will also receive rosuvastatin.

Nirmatrelvir/ritonavir will be given by mouth at the study clinic 2 times a day. Rosuvastatin will be given by mouth at the study clinic once (as a single dose).

We will compare participant experiences to help us determine the effect of nirmatrelvir/ritonavir on the pharmacokinetics of rosuvastatin.

Participants will take part in this study for approximately 11 weeks. During this time, they will have 10 days at the study clinic and 1 follow-up phone call. Blood samples will be collected during participants' time at the study clinic.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* BMI of 16-32 kg/m2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

* Positive test result for SARS-CoV-2 infection on Day -1.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinically relevant abnormalities requiring treatment (eg, acute myocardial infarction, unstable ischemic conditions, evidence of ventricular dysfunction, serious tachy or brady arrhythmias) or indicating serious underlying heart disease (eg, prolonged PR interval, cardiomyopathy, heart failure greater than NYHA 1, underlying structural heart disease, Wolff Parkinson-White syndrome).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Participants who have received a COVID-19 vaccine within 7 days before screening or admission, or who are to be vaccinated with a COVID-19 vaccine at any time during the study confinement period.
* A positive urine drug test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671052

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 healthy male and/or female participants were enrolled in the study.
Groups:
- Rosuvastatin Then Rosuvastatin + Nirmatrelvir/ Ritonavir: Period 1: Participants received a single oral dose of rosuvastatin 10 milligram (mg) on Day 1 of Period 1 in the morning (AM dose). Period 1 was followed by Period 2. Period 2: Participants received nirmatrelvir 100 mg and ritonavir 100 mg every 12 hours (BID) for 2 days (Day 1 of Period 2: morning [AM] and evening [PM]; Day 2 of Period 2: morning [AM]; total 3 doses) along with a single oral administration of rosuvastatin 10 mg on Day 2 of Period 2 in the morning (AM dose). Participants were followed-up to a maximum of 35 days from final dose of study intervention.
Period: Treatment Period 1 (Day -1 up to Day 5)
Arm/Group | Rosuvastatin Then Rosuvastatin + Nirmatrelvir/ Ritonavir
Started | 12
Completed | 12
Not Completed | 0
Period: Treatment Period 2 (Day 1 up to Day 5)
Arm/Group | Rosuvastatin Then Rosuvastatin + Nirmatrelvir/ Ritonavir
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who took at least 1 dose of study intervention.
Arm/Group | Rosuvastatin Then Rosuvastatin + Nirmatrelvir/ Ritonavir
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.75 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero (0) Extrapolated to Infinity (AUCinf) of Rosuvastatin in Period 1 and 2
Time Frame: Period 1: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1; Period 2: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post dose on Day 2
Population: Pharmacokinetic (PK) parameter set included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported. Here, "Number of Participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Groups:
- Period 1: Rosuvastatin 10 mg: Participants received a single dose of rosuvastatin 10 mg on Day 1 of Period 1 in the morning.
- Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg: Participants received nirmatrelvir 300 mg and ritonavir 100 mg BID for 2 days (Day 1 of Period 2: morning and evening and Day 2 of Period 2: morning, total 3 doses) along with a single oral administration of rosuvastatin 10 mg on Day 2 of Period 2 in the morning.
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
Number analyzed (Participants) | 11 | 11
Nanogram*hour per milliliter | 58.62 (46) | 72.78 (48)
Statistical Analysis 1: Comparison: Period 1: Rosuvastatin 10 mg vs Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg; Analysis was performed using mixed effect model with treatment as a fixed effect and participant within sequence as a random effect. Ratio of adjusted geometric means of test to reference was reported; where test treatment is Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg and reference treatment is Rosuvastatin 10 mg. Ratio and associated 90% CIs were reported in percentage; Test type: Other; Ratio of adjusted geometric means = 131.18, 90% CI 2-sided [115.89 to 148.48]

2. Primary Outcome: Maximum Observed Concentration (Cmax) of Rosuvastatin in Period 1 and 2
Time Frame: as for outcome 1
Population: PK parameter set included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
Number analyzed (Participants) | 12 | 12
Nanogram per milliliter | 5.691 (66) | 12.09 (60)
Statistical Analysis 1: Comparison: Period 1: Rosuvastatin 10 mg vs Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means = 212.44, 90% CI 2-sided [174.31 to 258.90]

3. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Rosuvastatin in Period 1 and 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
Number analyzed (Participants) | 12 | 12
Nanogram*hour per milliliter | 51.27 (61) | 71.13 (47)

4. Secondary Outcome: Time for Cmax (Tmax) of Rosuvastatin in Period 1 and 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
Number analyzed (Participants) | 12 | 12
Hours | 5.00 [3.00 to 5.10] | 2.00 [1.00 to 5.00]

5. Secondary Outcome: Terminal Half-Life (t1/2) of Rosuvastatin in Period 1 and 2
Description: t1/2 was calculated as loge (2) per kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 1
Population: PK parameter set included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported. Here, "Number of Participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
Number analyzed (Participants) | 11 | 11
Hours | 16.37 (6.0655) | 24.69 (8.2690)

6. Secondary Outcome: Apparent Clearance (CL/F) of Rosuvastatin in Period 1 and 2
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
Number analyzed (Participants) | 11 | 11
Liter per hour | 170.6 (46) | 137.4 (48)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Rosuvastatin in Period 1 and 2
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
Number analyzed (Participants) | 11 | 11
Liter | 3828 (53) | 4685 (59)

8. Secondary Outcome: Number of Participants With Clinically Significant Findings in Vital Signs
Description: Vital signs included blood pressure, pulse rate and temperature. Temperature was measured by orally. Blood pressure was measured with the participant in a supine position after 5 minutes of rest for the participant. Clinically significant findings were determined by the investigator.
Time Frame: Days 1 and 3 of each period
Population: Safety analysis set included all participants who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
Number analyzed (Participants) | 12 | 12
Participants
  Day 1 | 0 | 0
  Day 3 | 0 | 0

9. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory abnormalities criteria: a) Hematology: monocytes >1.2* upper limit of normal (ULN); b) Urinalysis: urine hemoglobin were >=1 and leukocyte esterase were >=1.
Time Frame: Day 1 of dosing up to 35 days up to last dose of study intervention (maximum of 45 days)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
Number analyzed (Participants) | 12 | 12
Participants | 4 | 2

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-emergent are events between first dose of study drug and up to 35 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 1 of dosing up to 35 days up to last dose of study intervention (maximum of 45 days)
Population: Safety analysis set consisted of all participants who received at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
Number analyzed (Participants) | 12 | 12
Participants | 5 | 10

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to 35 days up to last dose of study intervention (maximum of 45 days)
Arm/Group | Period 1: Rosuvastatin 10 mg | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Rosuvastatin 10 mg (N=12) | Period 2: Rosuvastatin 10 mg + Nirmatrelvir 300 mg/ Ritonavir 100 mg (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 10
Headache (Nervous system disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT05898672/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT05898672/SAP_001.pdf